CLINICAL TRIAL: NCT07382076
Title: Clinical Evaluation of the i-STAT ACTpro Cartridge Using Venous and Arterial Whole Blood Specimens on the i-STAT 1 Analyzer in an Adult Population
Brief Title: Clinical Evaluation of the i-STAT ACTpro Cartridge in an Adult Population
Acronym: ACT
Status: Active, not recruiting | Type: Observational
Sponsor: Abbott Point of Care (Industry)
Responsible Party: Sponsor
Other Study IDs: CS-2022-0009
Record Dates: First submitted 2026-01-26; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Activated Clotting Time
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Activated Clotting Time (ACT) in venous and arterial whole blood specimens.: Arterial and/or venous specimens from enrolled subjects will be tested in duplicate on the i-STAT 1 analyzer with the i-STAT ACTpro cartridge, and on the comparator device.
  Interventions: Diagnostic Test: Blood draw

INTERVENTIONS:
Diagnostic Test: Blood draw — A total volume of no more than 5mL of blood will be prospectively collected from subjects.

SUMMARY:
Measuring Activated Clotting Time (ACT) using the i-STAT ACTpro cartridge on the i-STAT 1 analyzer compared to a comparator device.

DETAILED DESCRIPTION:
The purpose of this study is to conduct a clinical evaluation of the investigational i-STAT ACTpro cartridge on the i-STAT 1 analyzer compared to a comparator device for measuring Activated Clotting Time (ACT) on venous and arterial whole blood specimens from adult participants.

The study will be conducted using whole blood specimens from participants undergoing Dialysis, Extracorporeal Life Support (ECLS)/ Extracorporeal Membrane Oxygenation (ECMO), and procedures in Electrophysiology Laboratories (EP Labs), Cardiac Catheterization Laboratories (Cath Labs), Interventional Radiology (IR) Units, and Cardiovascular Operating Rooms (CVOR).

ELIGIBILITY:
Inclusion Criteria:

* Subject is prescribed unfractionated heparin (UFH) peri-procedurally in order to reduce the risk of blood clots.

OR

- Subject for which only the baseline specimen (prior to UFH administration) is collected, subject is admitted for a medical procedure that would or could typically necessitate the use of UFH to reduce the risk of blood clots.

Exclusion Criteria:

* Prior enrollment in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults undergoing procedures where venous and arterial whole blood specimens are obtained in different care settings.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Compare ACT test results obtained from two different diagnostic devices. | Approximately thirty (30) to sixty (60) minutes depending on the length of the participants procedure and the number of research blood draws.
  Compare ACT test results obtained from the ACTpro cartridge using the i-STAT 1 analyzer with the ACT test result obtained from a comparator device using whole blood specimens.

SECONDARY OUTCOMES:
Precision assessment. | Approximately thirty (30) to sixty (60) minutes depending on the length of the participants procedure and the number of research blood draws.
  Conduct an assessment of precision for the ACT test using duplicate results generated using the i-STAT ACTpro cartridge on the i-STAT 1 analyzer.

CONTACTS AND LOCATIONS:
Overall Officials: Manish Gupta, MS, MBA, Study Director — Abbott Point of Care
Locations (11):
- United States (11):
  - Dignity Health Chandler Regional Medical Center, Chandler, Arizona
  - University of California at San Francisco, San Francisco, California
  - George Washington University, Washington D.C., District of Columbia
  - Kentucky Clinical Trials Laboratory, Louisville, Kentucky
  - University of Maryland, Baltimore, Maryland
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Penn State University Hershey Medical Center, Hershey, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Eastside Research Associates - Redmond, Redmond, Washington

IPD SHARING:
Plan to Share IPD: No